CLINICAL TRIAL: NCT06107816
Title: A Pilot, 3-arm Randomized Controlled Trial of a Fruit and Vegetable Prescription Program for Patients With Type Two Diabetes
Brief Title: A Fruit and Vegetable Prescription Program
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Susan Veldheer, Assistant Professor of Family and Community Medicine, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 23681; R01DK132077-01A1 (NIH)
Record Dates: First submitted 2023-10-16; First posted 2023-10-30 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Diabetes Mellitus; Diabetes Complications
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Complications

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual Care Control Group (Placebo Comparator): Will receive usual care
  Interventions: Behavioral: Usual Care
- F&V Rx Alone Group (Active Comparator): Will receive 4 monthly F&V Rx vouchers regardless of their DSME/S attendance.
  Interventions: Behavioral: F&V Rx alone
- F&V Rx + DSME/S Group (Active Comparator): Will receive monthly F&V Rx vouchers starting at the first group session and they will receive additional F&V Rx vouchers only when they attend a monthly DSME/S group (up to 4 total)
  Interventions: Behavioral: F&V Rx plus DSME/S

INTERVENTIONS:
Behavioral: Usual Care — Visit with a primary care provider and referral for diabetes self-management education and support (DSME/S) sessions
  Arms: Usual Care Control Group
Behavioral: F&V Rx alone — Usual Care plus four F&V prescriptions that are independent of DSME/S attendance
  Arms: F&V Rx Alone Group
Behavioral: F&V Rx plus DSME/S — Usual Care plus four F&V prescriptions that are dependent on DSME/S attendance
  Arms: F&V Rx + DSME/S Group

SUMMARY:
Dietary intake of fruits and vegetables (F&V) is a cornerstone for the treatment of type 2 diabetes, however less than 16% of Hispanic adults consume the recommended number of servings each day. F&V prescription (F&V Rx) programs are embedded into clinical settings and provide patients with vouchers to purchase F&V at local retailers. The proposed study aims to test the effects of a F&V Rx on diabetes self-management education and support (DSME/S) uptake and retention, dietary intake of F&V and diet quality, glucose control (hemoglobin A1c), and program implementation outcomes.

DETAILED DESCRIPTION:
Consuming a nutrient-dense diet, rich in fruits and vegetables (F&Vs) is at the cornerstone of type 2 diabetes (T2DM) treatment. Yet, among Hispanic adults, only 16% meet the recommended minimum F&V intake recommendations and have higher rates of T2DM than non-Hispanic whites (16.6% versus 13.3%, respectively). F&V Prescription (F&V Rx) programs are embedded in clinical settings, target medically high-risk patients such as those with T2DM, and provide them with vouchers to purchase F&V at local retailers. Preliminary F&V Rx studies in patients with T2DM have found F&V intake increases of 0.2-1.6 servings per day and hemoglobin A1c (A1c) reductions from 0.35-0.71% [3.8 -7.8 mmol/mol]. However, none of these studies included diabetes self-management education and support (DSME/S) which can lead to A1c decreases from 0.24% to 1.0% [2.6-10.9 mmol/mol]. The team conducted a pilot F&V Rx study where DSME/S attendance was incentivized by providing a F&V Rx at each session. Although DSME/S uptake is typically very low after referral (around 5-7%), the program had a 73% first session attendance rate. Further, at 7 months post-program, a clinically- and statistically-significant reduction was found in A1c of 1.3% [14.2 mmol/mol] (p=.001). Although the receipt of the F&V Rx vouchers was contingent upon DSME/S attendance in the study, other T2DM-focused F&V Rx studies did not have DSME/S attendance requirements and also saw A1c reductions. Thus, understanding the effect of a F&V Rx on DSME/S uptake and retention with and without attendance requirements is a key design issue that must be evaluated. This proposal is in response to PAS 20-160 for short-term, pilot randomized controlled trials (RCTs) to acquire preliminary data regarding trial design. The team proposes a 3-Arm, 16-week, pilot RCT (n=120) for low-income adults (aged 18+) with T2DM (A1c >7% [53 mmol/mol]). The control group (n=40) will receive usual care (UC). The two intervention groups (n=40 each) will receive UC plus a F&V Rx that is either independent of DSME/S attendance (F&V Rx alone) or dependent on DSME/S attendance (F&V Rx + DSME/S). First, the investigators will systematically explore the impact of a F&V Rx on uptake and retention in DSME/S. Next, the investigators will explore changes in A1c, and diet-related outcomes. Finally, with implementation in mind, the investigators will use Proctor's implementation taxonomy, and the cultural adaptation framework from Castro et al., to assess program appropriateness, acceptability, and sustainability with both participants and clinical care providers. The study team and the Community Advisory Board (CAB) have the research, clinical expertise, and established retail network necessary to conduct a F&V Rx trial in a low-income, Hispanic community. The findings of this trial will inform the design of a future, fully powered RCT and address gaps in knowledge related to how F&V Rx programs impact T2DM-related outcomes. If effective, F&V Rx programs have the potential to improve diabetes self-management and reduce the clinical burden of poor glycemic control, particularly in low-income, Hispanic communities.

ELIGIBILITY:
Inclusion Criteria:

* Patient at Penn State Health St. Joe's Medical Center
* Diagnosis of Type 2 Diabetes Mellitus greater than or equal to six months
* A1c level is greater than or equal to 7% (53 mmol/mol)
* Low income defined as enrolled in Supplemental Nutrition Assistance Program (SNAP), is uninsured or have Medicaid, or identifying as food insecure based on USDA criteria.
* Ability to give a blood sample
* Willing to respond to contacts from study staff over the study period
* Willing and able to give informed consent
* Can read and write in English or Spanish

Exclusion Criteria:

* Diagnosis of Type 2 Diabetes Mellitus less than six months
* Patients who have previously participated in the Veggie Rx program in the past year
* Patients who have attended any diabetes self-management education and support (DSME/S) sessions in the past year
* Women who are pregnant or who plan to become pregnant during the study period
* Any uncontrolled mental illness or substance abuse, or inpatient treatment for these in the past six months
* Any unstable or significant medical condition in the past 3 months (e.g. recent heart attack, stroke, DVT)
* A1c level is less than 7%
* Does not speak English or Spanish
* Inability to provide informed consent
* Unable to give a blood sample

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-07-26 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Evaluate the impact of a F&V Rx on DSME/S uptake in low-income adults | Throughout the 16 week intervention
  Defined as the number of participants who attend any 1 DSME (# attend any 1 DSME/S session/total # randomized)
Evaluate the impact of a F&V Rx on DSME/S retention in low-income adults. | Throughout the 16 week intervention
  Defined as % who attend >=75% of sessions (# attend >= 75% sessions/ # attended any 1 DSME/S session)

SECONDARY OUTCOMES:
Evaluate the impact of a F&V Rx on A1c (% and mg/dL) | Baseline (week 0) and follow up (week 16)
  Blood biomarker assessment will be taken and analyzed by the Penn State Health Clinical Labs.
Evaluate the impact of a F&V Rx on Diabetes Self-Management | Baseline (week 0) and follow up (week 16)
  Measured by DSME questionnaire
Evaluate the impact of a F&V Rx on Fruit and Vegetable Intake | Baseline (week 0) and follow up (week 16)
  Based on the 24-hour recalls
Evaluate the impact of a F&V Rx on Healthy Eating index-2015 | Baseline (week 0) and follow up (week 16)
  Based on the 24-hour recalls
Evaluate the impact of a F&V Rx on Total plasma carotenoids (ng/mL) | Baseline (week 0) and follow up (week 16)
  Plasma carotenoids will be separated into the total and five individual concentrations (α-carotene, β-carotene, lutein, lycopene, and cryptoxanthin) using high-performance liquid chromatography methodology using our Sciex Exion LC-Sciex QTRAP 6500+ mass spectrometry system.
Evaluate the impact of a F&V Rx on Food insecurity | Baseline (week 0) and follow up (week 16)
  Measured by the 18-item USDA Food Insecurity Questionnaire

OTHER OUTCOMES:
Assess program implementation outcomes - Acceptability of Intervention Measure (AIM) | Throughout the 16 week intervention and follow-up
  A four-item measure implementation outcomes to assess acceptability of the DSME/S sessions and the overall intervention for participants.
Assess program implementation outcomes - Intervention Appropriateness Measure (IAM) | Throughout the 16 week intervention and follow-up
  A four-item measure of implementation to assess the appropriateness of the DSME/S sessions and the overall intervention for participants.
Assess program implementation outcomes - Clinic/providers/staff - Implementation Outcomes Questionnaire (IOQ) | Throughout the 16 week intervention and follow-up
  Survey that measures implementation success of the intervention from the perspective of stakeholders who carry out the daily operations

CONTACTS AND LOCATIONS:
Overall Officials: Susan Veldheer, DEd, RD, Principal Investigator — Penn State College of Medicine
Locations (1):
- Penn State Health St. Joseph Downtown Campus, Reading, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No